CLINICAL TRIAL: NCT02113007
Title: Phase II Study of High-Dose Rituximab Combined With Temozolomide as Treatment for Patients With Primary CNS Lymphoma
Brief Title: Study of High-Dose Rituximab With Temozolomide as Treatment for Primary Central Nervous System (CNS) Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed early due to slow accrual.
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI CNS 20
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Lymphoma; CNS; rituximab; temozolomide
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab plus Temozolomide (Experimental): Rituximab: 375 mg/m2 IV, days 1, 3, and 5 Temozolomide: 150 mg/m2 PO, days 1-5
  Interventions: Drug: Rituximab plus Temozolomide

INTERVENTIONS:
Drug: Rituximab plus Temozolomide — Treatment cycles will be repeated every 14 days (2 weeks) for the lead-in portion. If no prohibitive toxicities are observed in the first 6 patients during the first 2 treatment cycles, the study will continue enrolling patients. Treatment cycles for the Phase II portion will be repeated every 14 days (2 weeks) for a total of 12 cycles.
  Other Names: Rituximab: Rituxin, MabThera; Temozolomide: Temodar

SUMMARY:
This study will evaluate the safety and efficacy of high-dose rituximab combined with temozolomide in the treatment of patients with Primary Central Nervous System Lymphomas (PCNSL). This novel combination will be evaluated in PCNSL patients who are 60 years of age or older, or in patients 18 years or older who refuse methotrexate-based treatment.

DETAILED DESCRIPTION:
This is a Phase II, multi-centered, single-arm study. A brief patient lead-in portion will be included to assess safety and feasibility. The first six patients enrolled will be monitored weekly for safety during two treatment cycles (4 weeks) for adverse events to assure there are no unexpected or prohibitive toxicities. If safety signals emerge from this group of patients, the protocol may be discontinued or modified.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed CD20 positive primary B-cell CNS lymphoma (PCNSL) confirmed by one of the following:

   * Brain biopsy or resection;
   * Cerebrospinal fluid (CSF) cytology for lymphoma or monoclonal lymphocyte population as defined by cell surface markers.
2. No evidence of systemic non-Hodgkin's lymphoma.
3. Male or female, and:

   * 60 years of age or older, or
   * 18 years of age or older and decline methotrexate-based treatment.
4. Measurable contrast-enhancing disease by MRI of brain and or spine (with gadolinium contrast).
5. ECOG PS equals 2 or less.
6. No more than 2 prior chemotherapy regimens.
7. Adequate hematologic, renal, and hepatic function.
8. Ability to swallow oral medications.
9. Female patients who are not of childbearing potential, and female patients of childbearing potential who agree to use adequate contraceptive measures, who are not breastfeeding, and who have a negative serum pregnancy test within 72 hours prior to start of treatment.
10. Male patients willing to use adequate contraceptive measures.
11. Life expectancy 8 weeks or greater.
12. HIV negative.
13. Archival tumor block (or 20 unstained slides) for biomarker testing. Patients without archived tumor block material will be allowed to participate in the study.
14. Willingness and ability to comply with study and followup procedures.
15. Ability to understand the nature of this study and give written informed consent.
16. Bone marrow biopsy must be negative for lymphoma.

Exclusion Criteria:

1. Previous treatment with rituximab or other monoclonal antibodies, or temozolomide.
2. Prior bone marrow or organ transplantation.
3. Chemotherapy or investigational drug therapy for cancer up to 21 days prior to day-1 of study.
4. T-cell primary CNS lymphoma.
5. Known hypersensitivity to dacarbazine (DTIC).
6. Active, clinically serious infection greater than CTCAE grade 2. Patients may be eligible upon resolution of the infection.
7. Positive test results for chronic hepatitis BsAg infection.
8. Chronic treatment with steroids or other immunosuppressive agents for medical conditions other than cancer. Patients who require steroids for treatment of tumor-associated cerebral edema are eligible.
9. History of other malignancy up to 5 years prior to study entry which could affect compliance with the protocol or interpretation of results. History of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix, low grade, early stage, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ (DCIS) of the breast treated with lumpectomy alone with curative intent, are generally eligible.
10. History of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment), New York Heart Association Classification III or IV.
11. Vaccination with a live-virus vaccine up to 4 weeks prior to onset of study treatment.
12. Impairment of gastrointestinal (GI) function or GI disease that, in the opinion of the investigator, may significantly alter the absorption of study drug (e.g., Crohn's disease, ulcerative disease, uncontrolled vomiting, diarrhea, or malabsorption syndrome).
13. Significant, concurrent, uncontrolled medical condition which, in the opinion of the investigator, may interfere with patient participation in the study.
14. Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Shih, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (4):
- United States (4):
  - Yale School of Medicine, New Haven, Connecticut
  - Memorial Cancer Institute, Hollywood, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Tennessee Oncology PLLC, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In August 2015, 2 patients with confirmed primary central nervous system (CNS) lymphoma were enrolled in the trial. Only one (of 4) investigational sites in the U.S accrued patients. Due to slow enrollment, the study was terminated in February 2016.
Period: Overall Study
Arm/Group | Rituximab Plus Temozolomide
Started | 2
Completed | 0
Not Completed | 2
Not completed — Progressive disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab Plus Temozolomide
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Patients will be assessed for response by MRI of brain and/or spine after 4 cycles (8 weeks) of treatment according to Response Criteria for Primary CNS Lymphoma. Patients with stable disease or better (CR or PR) will continue treatment for 12 cycles (24 weeks). Complete Response (CR)=no contrast enhancement, normal eye exam. Partial Response (PR)=50 percent decrease in tumor enhancement, minor retinal pigment epithelium abnormality in eye exam. Stable disease (SD)= a change in lesion size that is neither sufficient shrinkage to qualify for a PR nor sufficient increase to qualify for progressive disease.
Time Frame: approximately 32 weeks
Population: The study closed early due to slow accrual. This outcome measure was not reached.
Arm/Group | Rituximab Plus Temozolomide
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Six and twelve-month CNS progression-free survival rate.
Time Frame: 6 and 12 months
Population: The study closed early due to slow accrual; outcome measure not reached.
Arm/Group | Rituximab Plus Temozolomide
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events as a Measure of Safety.
Description: Patients in the safety lead-in part of the study were monitored for up to 2 treatment cycles (4 weeks) to assure there were no unexpected or prohibitive toxicities. A non-serious adverse event is any untoward medical occurrence. A serious adverse event (SAE) is an event that meets one or more of the following: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; requires intervention to prevent permanent impairment or damage. Specific AE and SAE terms are provided in the Adverse event module.
Time Frame: up to 4 weeks
Measure: Number; unit: participants
Arm/Group | Rituximab Plus Temozolomide
Number analyzed (Participants) | 2
participants
  Adverse Events | 2
  Serious Adverse Events | 1

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for up to 4 weeks during the safety lead-in part of the study. The study closed early due to slow accrual.
Arm/Group | Rituximab Plus Temozolomide
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Plus Temozolomide (N=2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Plus Temozolomide (N=2)
Flatulence (Gastrointestinal disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Gait disturbance (General disorders) | 1
Fatigue (General disorders) | 2

LIMITATIONS AND CAVEATS:
Two (2) subjects were enrolled in the safety lead-in part of the study. The study closed early due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.